CLINICAL TRIAL: NCT07348991
Title: Predicting Atrial Fibrillation and Life-threatening Cardiac Arrhythmias and Conduction Disorders in the Perioperative Period in High Cardiac Risk Surgery Using Artificial Intelligence Elements
Brief Title: Predicting Severe Cardiac Arrhythmias in the Perioperative Period Using AI-ECG
Status: Not yet recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ChPSH1
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation; Atrioventricular Block, Second and Third Degree; Sinus Node Dysfunction; Ventricular Tachycardia (VT); Ventricular Fibrillation
Keywords: Electrocardiogram; Artificial intelligence; Cardiac arrhythmias; Atrioventricular block; Perioperative; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Atrioventricular Block; Neoplasm Metastasis; Sick Sinus Syndrome; Tachycardia, Ventricular; Ventricular Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention group: patients meeting the inclusion criteria who are hospitalised for surgery with a high cardiovascular risk
  Interventions: Diagnostic Test: digital single-channel ECG recording

INTERVENTIONS:
Diagnostic Test: digital single-channel ECG recording — A single-channel ECG will be recorded for 3 minutes while the patient is sitting at rest. The patient leans back against the chair, legs uncrossed, and arms resting on the knees or on the table. Standard lead I is recorded using the CardioQVARK software and hardware complex (CardioQVARK medical device (Electrocardiograph) issued by Roszdravnadzor (Federal Service for Surveillance in Healthcare) P3H 2024/22855, issued on June 5, 2024).

SUMMARY:
During the preoperative examination, in addition to the standard examination recommended before high-risk cardiac surgeries, a digital single-lead ECG is recorded using portable CardioQUARK devices. This ECG is analyzed for time, amplitude, and frequency parameters-more than 200 parameters per cardiac cycle. Additionally, the available parameters of a standard 12-lead ECG recording are determined. All parameters of both single-lead and 12-lead ECGs will be included in a multivariate regression analysis to determine the optimal method for predicting atrial fibrillation, life-threatening cardiac arrhythmias, and conduction abnormalities in the perioperative period after high-risk cardiac procedures.

The study will include patients undergoing high-risk cardiac surgeries, such as those on the heart, aorta, esophagus, pancreas, liver, and lungs, as well as high-risk oncological surgeries. A partial analysis will also be performed depending on the type of intervention. Rhythm and conduction disturbances will be recorded during surgery, as well as in the postoperative period, using ECG monitors, 24-hour ECG monitoring, and repeated recordings of a standard ECG when complaints or signs of unstable hemodynamics arise

DETAILED DESCRIPTION:
In study, the investigators plan to identify single-channel and 12-lead ECG parameters that correlate significantly with the occurrence of atrial fibrillation and life-threatening cardiac arrhythmias and conduction disturbances in the perioperative period after high-risk cardiac interventions.

A prospective, non-randomized, observational, controlled, single-center study consisting of two consecutive stages is being conducted.

The first stage involves identifying single-channel and 12-lead ECG parameters that correlate significantly with the onset of atrial fibrillation and life-threatening cardiac arrhythmias and conduction disorders in the perioperative period after interventions with high cardiac risk. Participants who meet the inclusion criteria will undergo the following during preoperative preparation: recording of a digital single-channel ECG using the CardioQVARK software and hardware complex (CardioQVARK medical device (Electrocardiograph) issued by Roszdravnadzor (Federal Service for Surveillance in Healthcare) P3H 2024/22855, issued on June 5, 2024); a digital 12-lead ECG; an extended echocardiographic examination; and 24-hour Holter ECG monitoring.

The single-channel ECG will be recorded for 3 minutes at rest in a sitting position. The participants leans back against the back of the chair, legs uncrossed, arms resting on the knees or on the table. Standard lead I is recorded using the CardioQVARK software and hardware complex.

Next, the parameters of single-channel and 12-channel ECG are identified that have a reliable correlation with the occurrence of atrial fibrillation and life-threatening arrhythmias and conduction disorders in the perioperative period after interventions with high cardiac risk, followed by the creation of a machine learning model and/or or neural network analysis with deep learning support for predicting the occurrence of atrial fibrillation and life-threatening arrhythmias and conduction disorders.

The second stage will involve testing using a test sample of the algorithm, taking into account the ECG parameters which, according to the statistical analysis performed in the first stage, had the highest sensitivity and specificity in predicting the onset of atrial fibrillation and life-threatening cardiac arrhythmias and conductions disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age;
* Scheduled surgery with high cardiac risk
* Informed consent was given to participate in the study

Exclusion Criteria:

* Cancellation of the surgery for any reason;
* The patient's unwillingness to continue participating in the study;
* Poor quality of the ECG recording on a single-channel ECG monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will analyze patients undergoing elective high-risk cardiac surgeries, including cardiac surgery, aortic surgery, esophageal and gastric cardia surgery, and thoracic surgery. Patients undergoing large-scale oncological surgeries will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
specificity, sensitivity, prognostic significance of a positive and negative result, diagnostic accuracy | 30 days after sugery starts
  statistical parameter of diagnostic and prognostic accuracy of the method under study
specificity, sensitivity, prognostic significance of a positive and negative result, prognostic significance of a positive and positive result, diagnostic accuracy | perioperative period - from the surgery starts till 30 days after surgery
  statistical parameter of diagnostic and prognostic accuracy of the method under study

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 01.2026-01.2028
Access Criteria: email call

REFERENCES:
- [Background] Paroxysms of atrial fibrillation during planned cardiac surgery under artificial circulation / E. P. Gulyaeva-Seltsovskaya, I. Dkhif, A. A. Mols [et al.] // Bulletin of the Smolensk State Medical Academy. - 2023. - Vol. 22, No. 4. - P. 100-106. - DOI 10.37903/vsgma.2023.4.14. - EDN MIIWSU
- [Background] Chomakhidze P.Sh., Kurbanalieva N.K., Nebezhev A.A., Sedov V.P., Syrkin A.L. Modern aspects of preoperative examination in planned extracardiac interventions. Consilium Medicum. 2025;27(1): DOI: 10.26442/20751753.2025.1.203060 © CONSILIUM MEDICUM LLC, 2025